CLINICAL TRIAL: NCT05208086
Title: Diagnostic Performance of Spot Urine Sample for the Monoclonal Components Detection in Patients With Multiple Myeloma RHU(M)M Random or H24 Urine in (Multiple) Myeloma
Brief Title: Diagnostic Performance of Spot Urine Sample for the Monoclonal Components Detection in Patients With Multiple Myeloma
Acronym: RHUMM
Status: Recruiting | Type: Observational
Sponsor: Intergroupe Francophone du Myelome (Network)
Responsible Party: Sponsor
Other Study IDs: IFM 2020-03
Record Dates: First submitted 2021-12-16; First posted 2022-01-26 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Monoclonal components detection; Urine sample
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Cycle1 day1: collection of 24h urine and an urine sample from miction the day of the visit.
  Cycle 2 day1:collection of 24h urine and an urine sample from miction the day of the visit Cycle 4 day 1: collection of 24h urine and an urine sample from miction the day of the visit.
  Interventions: Diagnostic Test: Detection of monoclonal component

INTERVENTIONS:
Diagnostic Test: Detection of monoclonal component — Monoclonal component analysis by electrophoresis and immnuofixation on the urine sample from miction and 24h urine sample.

SUMMARY:
The primary objective of the study is to evaluate at Day 1 Cycle 2, the detection sensitivity of the urinary monoclonal component on a spot urine sample, compared to the reference measurement on 24-hour urine, in patients with Multiple Myeloma.

DETAILED DESCRIPTION:
To evaluate the detection sensitivity of the urinary monoclonal component on a spot urine sample, compared to the reference measurement on 24-hour urine, in Multiple Myeloma patients.

300 evaluable patients are required. For each of them, both spot urine sample and 24h urine sample will be collected at Cycle1 Day1, Cycle 2 Day 1 and Cycle 4 Day 1.

The detection of urine monoclonal component will be performed by urine protein electrophoresis (quantitative) and urine immunofixation (qualitative).

ELIGIBILITY:
Inclusion Criteria:

* Patient with Multiple Myeloma
* Patient starting new treatment line, whatever the line is, but with at least 3 induction cycles
* Urine monoclonal component ≥ 200mg/24h

Exclusion Criteria:

Person under guardianship, trusteeship or deprived of freedom by a judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Multiple Myeloma whatever the line of treatment started in one of the twenty investigators sites located in France.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Evaluate the detection sensitivity of the urine monoclonal component on spot urine sample | at the first Day of Cycle n°2 (each cycle is 28 days or 21 days)
  Evaluate the detection sensitivity of the urine monoclonal component on spot urine sample compared to the reference measurement of 24 hours urine.
  Sensitivity is defined as the proportion, among the patients with positive urinalysis results on 24 hours urine, of positive results on spot urine sample. Evaluation is performed by urine protein electrophoresis and urine immunofixation

SECONDARY OUTCOMES:
Evaluate the specificity of urine monoclonal component detection on spot urine sample | at the first Day of cycle n°2 (each cycle is 28 days or 21 days)
  Evaluate the specificity of urine monoclonal component detection on sample at C2D1 compared to the reference measurement of 24 hours urine sample.
  Specificity is defined as the proportion, among patients with negative urinalysis results on 24 hours urine, of negative results on the spot urine sample.
Evaluate the sensitivity and specificity of urine monoclonal component detection on spot urine sample | at the first day of cycle n°1 and cycle n°4 (each cycle is 28 days or 21 days)
  Evaluate the sensitivity and specificity of urine monoclonal component detection on spot urine sample at C1D1 and C4D1 compared to reference measurement of 24hours urine sample
Compare the responses rate | at the first day of cycle n° 2 and cycle 4 (each cycle is 28 days or 21 days)
  Compare the rate of partial responses, very good partial responses and complete responses (IMWG criteria) but only on the urinary monoclonal component) at C2D1 and C4D1 between the two types of samples (spot urine sample and 24hours urine sample)
Compare the monoclonal component / creatininuria ratios | at the first day of cycle n° 1,2 and 4
  Compare the monoclonal component / creatininuria ratios in both samples (spot urine sample and 24hours urine sample) for components monoclonal which are quantifiable in both types of urine samples
Define the equivalent of 200 mg / 24H (current consensus threshold of measurable urinary disease) | at the first day of cycle n° 1 (each cycle is 28 days or 21 days)
  Define the equivalent of 200 mg / 24H (current consensus threshold of measurable urinary disease) at C1D1 and on the others points, if the monoclonal component is quantifiable)
Assess the association between the rate of serum light chains and concentration of monoclonal components | at first day of cycle 2 (each cycle is 28 days or 21 days)
  To assess the association between serum light chains and concentration of monoclonal components for both types of urine samples.
Evaluate the urine monoclonal component by the difference between proteinuria and albuminuria | at first day of cycle 2 (each cycle is 28 days or 21 days)
  To Evaluate if the rate of urine monoclonal component (in g/L)could by calculated by the difference between proteinuria (in g/L) and albuminuria (in g/L)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier DECAUX, PU-PH, Principal Investigator — Rennes University Hospital
Locations (20):
- France (20):
  - Ch Annecy Genevois, Annecy
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - Centre Hospitalier Métropole de Savoie, Chambéry
  - CHU François Mitterand, Dijon
  - CH de Dunkerque, Dunkirk
  - CHD Vendée, La Roche-sur-Yon
  - Hopital Bicètre, Le Kremlin Bicètre
  - Ch Le Mans, Le Mans
  - CH de Lens, Lens
  - Hopital Claude Huriez-CHRU LILLE, Lille
  - Centre Hospitalier Lyon sud, Lyon
  - CHU de Montpellier, Montpellier
  - Hôpital E. MULLER, Mulhouse
  - CHRU Nantes, Nantes
  - CHU de Reims, Reims
  - Chu Pontchaillou, Rennes
  - CHU Toulouse, Toulouse
  - CHRU Bretonneau, Tours
  - CH Bretagne Atlantique Vannes et Auray-P.Chubert, Vannes
  - CH de Versailles, Versailles